CLINICAL TRIAL: NCT07058727
Title: The Effect of Different Hemostatic Agents Used in Partial Pulpotomy on Pulp Survival and Postoperative Pain: A Randomized Clinical Trial
Brief Title: Different Hemostatic Agents Used in Partial Pulpotomy on Pulp Survival and Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra SUSGUN YILDIRIM, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP-HemoRCT-2025
Record Dates: First submitted 2025-06-19; First posted 2025-07-10 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Efficacy of Hemostatic Agents; Partial Pulpotomy; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): 2.5% NaOCl applied for 1 min after pulp exposure.
  Interventions: Drug: Sodium Hypochlorite 2,5%
- Arm 2 (Experimental): 2% CHX applied for 1 min
  Interventions: Drug: Chlorhexidine
- Arm 3 (Experimental): Hemostasis achieved with 4°C saline for 1 min.
  Interventions: Drug: Cold Saline

INTERVENTIONS:
Drug: Sodium Hypochlorite 2,5% — 2.5% NaOCl applied for 1 min to exposed pulp for hemostasis, followed by standard pulp capping
  Arms: Arm 1
Drug: Chlorhexidine — 2% CHX applied for 1 min to achieve hemostasis, with identical subsequent steps to NaOCl group
  Arms: Arm 2
Drug: Cold Saline — Hemostasis via 4°C saline (1 Min), then standardized pulp capping
  Arms: Arm 3

SUMMARY:
This randomized clinical trial evaluates the efficacy of sodium hypochlorite (NaOCl), chlorhexidine (CHX), and cold saline as hemostatic agents in partial pulpotomy. The study compares postoperative pain (via VAS scores) and pulp survival (via clinical/radiographic evaluation) at 1, 3, 7 days, 6 months, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth with carious pulp exposure (no spontaneous pain).
* Positive vitality test (Endo-Ice).
* No periapical radiolucency.

Exclusion Criteria:

* Systemic diseases affecting healing.
* Pregnancy.
* Non-vital pulp/necrosis

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 1 week
  The patient will be asked to rate the pain on the 1st, 3rd and 7th day according to VAS. (The patient is asked to score their pain in this range, with 0 being the lowest and 10 being the highest.)
Pulp Survival Rate | 12 months
  The pulp is expected to be vital, without percussion tenderness and without spontaneous pain

SECONDARY OUTCOMES:
Clinical Success | 12 months
  Maintaining the integrity of the restoration No need for endodontics treatments